CLINICAL TRIAL: NCT06182111
Title: Intraoperative Administration of Intravenous Morphine in Patients Undergoing Laparoscopic Cholecystectomy - a Retrospective, Observational, Quality-improvement Study
Brief Title: Intraoperative Administration of Intravenous Morphine in Patients Undergoing Laparoscopic Cholecystectomy
Acronym: MORPHLAPCHOL
Status: Recruiting | Type: Observational
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Sanne Vibe Nielsen, Principal investigator, Esbjerg Hospital - University Hospital of Southern Denmark
Other Study IDs: 23/47526
Record Dates: First submitted 2023-11-14; First posted 2023-12-26 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Pain; Morphine; Laparoscopic Cholecystectomy
Keywords: Intraoperative morphine for laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No morphine: Participants who have undergone surgery before anesthesia protocol was changed. These participants have not received morphine during surgery.
- Morphine: Participants who have undergone surgery after anesthesia protocol was changed. These participants have received morphine during surgery.
  Interventions: Procedure: Intraoperative morphine

INTERVENTIONS:
Procedure: Intraoperative morphine — Morphine dose = 0,1 mg mg/kg (maximum 10 mg) intravenous given 20 min after start of surgery
  Groups: Morphine

SUMMARY:
The goal of this observational, quality improvement study is to compare the effect of a dose of morphine given during gall-bladder removal surgery. The main questions to answer are:

* Do participants, who are given given a dose of morphine during gall-bladder removal surgery, experience less pain after surgery?
* Does a dose of morphine during gall-bladder removal surgery cause more side effects? The investigators will compare the effects of two types of anesthesia: a) anesthesia without morphine during surgery, and b) anesthesia with morphine during surgery.

DETAILED DESCRIPTION:
The investigators will use Redcap secure web application (via Open Patient Data Explorative Network, a subsidiary under University Hospital of Odense, Denmark) for data collection and data management.

No sample size has been collected as per the observational design. The investigators expect to include an equal number in each study arm, as there has been no indication of change in indications for surgery type.

The investigators expect to use students T-test for comparison of groups. If possible logistic regression analyses will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* patients who have had elective laparoscopic cholecystectomy/planned gall-bladder removal surgery

Exclusion Criteria:

* age limit as above
* patients unable to give consent to anesthesia
* patients unable to participate in pain scoring
* patients with chronic pain syndromes, characterized by patients receiving regular analgesic treatment and patients with active or previous contact to pain clinic)
* patients with active or previous substance abuse
* emergency surgery

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Surgery performed at Hospital og South West Jutland, Esbjerg in main operating facilities.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Use of rescue analgesia. | 24 hours
  Calculated as morphine equivalents.

SECONDARY OUTCOMES:
Intraoperative opioid use. | 24 hours
  Calculated as morphine equivalents.
Pain-score at arrival in postoperative ward. | 24 hours
  Intervals: 0 = no pain, 1 = light pain (equivalent to numerical ranking scale (NRS) 1-3), 2 = moderate pain (equivalent to NRS 4-6), 3 = severe pain (equivalent to NRS 7-10).
Pain-score at discharge from postoperative ward. | 24 hours
  Intervals: 0 = no pain, 1 = light pain (equivalent to NRS 1-3), 2 = moderate pain (equivalent to NRS 4-6), 3 = severe pain (equivalent to NRS 7-10).
Rescue antiemetic treatment in postoperative ward. | Up to 24 hours follow up.
  Antiemetic drugs and doses registered.
Time in postoperative ward. | 24 hours
  Minutes.
Analgesic treatment in surgical ward if admitted | 24 hours
  Only if admitted (a large proportion of patients expected to undergo out-patient procedure). Calculated as morphine equivalents.
Antiemetic treatment in surgical ward. | 24 hours
  Only if admitted (a large proportion of patients are expected to undergo out-patient procedure). Antiemetic drugs and doses registered.
Hospital length of stay. | 1 month
  Only if admitted (a large proportion of patients are expected to undergo out-patient procedure).
Emergence from anesthesia. | 24 hours
  Surrogate measure of emergence from anesthesia time.

CONTACTS AND LOCATIONS:
Overall Officials: Sanne V Nielsen, MD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (1):
- Hospital of south West Jutland, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
At this time implications of answering in the affirmative are unknown, and description of shared individual participant data (IPD)s cannot be done yet.
  However, the investigators fully expect to share anonymized IPD in order to be able to publish the results ogf the study in a peer reviewed journal.

DOCUMENTS (1):
  • Study Protocol (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT06182111/Prot_000.pdf